CLINICAL TRIAL: NCT01154439
Title: A Phase I Study Investigating the Combination of RAD001 With Standard Induction and Consolidation Therapy in Older Patients With Newly Diagnosed Acute Myeloid Leukemia (AML)
Brief Title: Everolimus MICE-regimen in Treating Older Patients With Newly Diagnosed Acute Myeloid Leukemia
Acronym: AML1208
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gruppo Italiano Malattie EMatologiche dell'Adulto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AML1208; GIMEMA-AML1208 (Other: GIMEMA Foundation); 2008-007666-28 (EudraCT Number)
Record Dates: First submitted 2010-06-29; First posted 2010-06-30 (Estimated); Last update posted 2022-10-26 (Actual); Status verified 2022-10

CONDITIONS: Leukemia
Keywords: secondary acute myeloid leukemia; untreated adult acute myeloid leukemia; adult acute basophilic leukemia; adult acute eosinophilic leukemia; adult erythroleukemia (M6a); adult pure erythroid leukemia (M6b); adult acute megakaryoblastic leukemia (M7); adult acute minimally differentiated myeloid leukemia (M0); adult acute monoblastic leukemia (M5a); adult acute monocytic leukemia (M5b); adult acute myeloblastic leukemia with maturation (M2); adult acute myeloblastic leukemia without maturation (M1); adult acute myelomonocytic leukemia (M4); adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22)
MeSH Terms: conditions — Leukemia; Leukemia, Basophilic, Acute; Leukemia, Eosinophilic, Acute; Leukemia, Erythroblastic, Acute; Leukemia, Megakaryoblastic, Acute; Leukemia, Monocytic, Acute; Leukemia, Myeloid, Acute; Leukemia, Myelomonocytic, Acute; Congenital Abnormalities | interventions — Cytarabine; Idarubicin; Etoposide; Everolimus; Mitoxantrone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Everolimus (Experimental): Everolimus mice-regimen
  Interventions: Drug: cytarabine; Drug: etoposide; Drug: everolimus; Drug: idarubicin; Drug: mitoxantrone hydrochloride

INTERVENTIONS:
Drug: cytarabine — Remission induction therapy: by short i.v. infusion on days 1 and 7. Consolidation therapy: by continuous infusion on days 1-5.
  Other Names: Mini-ICE regimen (idarubicin, cytarabine and etoposide).
Drug: etoposide — Remission induction therapy: by short i.v. infusion, on days 1-7. Consolidation therapy: by short i.v. infusion, on days 1-5.
  Other Names: Mini-ICE regimen (idarubicin, cytarabine and etoposide).
Drug: everolimus — Remission induction therapy: test dose once a day by mouth, on days 1-21 (21 days).
  Consolidation therapy: dose as defined by the cohort once a day by mouth, on days 1-10.
  Other Names: RAD001
Drug: idarubicin — Consolidation therapy: by short infusion i.c. on days 1, 3 and 5.
  Other Names: Mini-ICE regimen (idarubicin, cytarabine and etoposide).
Drug: mitoxantrone hydrochloride — Remission induction therapy: by short i.v. infusion on days 1, 3 and 5

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as mitoxantrone hydrochloride, cytarabine, etoposide, and idarubicin, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Everolimus may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the cancer. Giving everolimus together with combination chemotherapy may kill more cancer cells.

PURPOSE: This phase I trial is studying the side effects and best dose of everolimus when given together with mitoxantrone hydrochloride, cytarabine, etoposide, and idarubicin in treating older patients with newly diagnosed acute myeloid leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the maximum-tolerated dose of everolimus in combination with standard remission-induction therapy comprising mitoxantrone hydrochloride, cytarabine, and etoposide (MICE-regimen) followed by consolidation therapy comprising idarubicin, cytarabine, and etoposide in older patients with newly diagnosed acute myeloid leukemia.

Secondary

* To determine the safety profile of this regimen in these patients.
* To determine the anti-leukemic activity (complete remission rate [complete remission and complete remission with incomplete blood count recovery]) following one or two induction courses.

OUTLINE: This is a multicenter, dose-escalation study of everolimus.

* Standard remission-induction therapy: Patients receive mitoxantrone hydrochloride IV over 30 minutes on days 1, 3, and 5; cytarabine IV continuously on days 1-7; etoposide IV over 1 hour on days 1-3; and oral everolimus once a day on days 1-21. Patients with partial remission (PR) receive a second induction course, beginning 7-17 days after completion of induction course 1. Patients with complete remission or complete remission with incomplete blood count recovery (CR/CRi) after induction therapy proceed to consolidation therapy; patients who have failed to achieve PR after induction course 1 or a CR/CRi after induction course 2 are removed from study.
* Consolidation therapy: Beginning within 3 weeks from CR/CRi documentation, patients receive idarubicin IV over 30 minutes on days 1, 3, and 5; cytarabine IV continuously on days 1-5; etoposide IV over 1 hour on days 1-3; and oral everolimus once a day on days 1-10. Patients may receive another course of the consolidation therapy, beginning at least 4 weeks after initiation of consolidation therapy course 1.

After completion of study treatment, patients are followed up once a month for 1 year, every 3 months for 1 year, and then periodically thereafter.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Newly diagnosed acute myeloid leukemia (AML) (unequivocal) according to WHO diagnostic criteria (at least 20% blasts in the bone marrow), with FAB classification other than M3 (acute promyelocytic leukemia), and documented by bone marrow aspiration (or biopsy in case of dry tap)
* Previously untreated primary or secondary AML (including AML following antecedent myelodysplasia)
* No blast transformation of chronic myeloid leukemia or other myeloproliferative disorders
* No active CNS leukemia

PATIENT CHARACTERISTICS:

* WHO performance status 0-2
* Total serum bilirubin < 2 times upper limit of normal (ULN)
* Serum creatinine < 2 times ULN
* ALT/AST ≤ 3 times ULN (unless due to organ leukemic involvement)
* LVEF ≥ 50% by echocardiogram
* No other concurrent active malignancy
* No active uncontrolled infection
* No known active hepatitis B or C or HIV positivity
* No active heart disease including myocardial infarction within the past 3 months, symptomatic coronary artery disease, cardiac arrhythmias not controlled by medications, or uncontrolled congestive heart failure
* No medical condition that, in the opinion of the investigator, places the patient at an unacceptably high risk for toxicities
* No other known condition (e.g., familial, sociological, or geographical) or behavior (including drug dependence or abuse, psychological or psychiatric illness) that, in the opinion of the investigator, would make the patient a poor candidate for the trial
* No known hypersensitivity to everolimus, other rapamycins (e.g., sirolimus or temsirolimus), or to its excipients

PRIOR CONCURRENT THERAPY:

* No prior standard or investigational chemotherapy for acute myeloid leukemia or myelodysplasia (including everolimus or other mTOR inhibitors)

  * Prior hydroxyurea allowed (up to a maximum of 14 days) to control peripheral blood leukemic cell counts
* No prior enrollment in this trial
* No other concurrent anti-leukemia agents, investigational agents, or biological agents

Ages: 61 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2010-10; Primary Completion 2013-05 (Actual); Study Completion 2015-09-15 (Actual)

PRIMARY OUTCOMES:
Maximum-tolerated dose of everolimus | At one year from study entry
  MTD of RAD given in combination with the MICE regimen

SECONDARY OUTCOMES:
Safety | At one year from study entry
Complete remission rate | At one year from study entry
  Complete remission rate (CR + CRi) following one or two induction courses.

CONTACTS AND LOCATIONS:
Overall Officials: Sergio Amadori, MD, Principal Investigator — Azienda Ospedaliera Universitaria Policlinico Tor Vergata
Locations (5):
- Italy (5):
  - Ematologia con trapianto- AOU Policlinico Consorziale di Bari, Bari
  - Azienda Ospedaliera Universitaria - Università degli Studi di Napoli "Federico II" - Facoltà di Medicina e Chirurgia, Napoli
  - Università La Sapienza, Roma
  - Università degli Studi "Sapienza" - Dip Biotecnologie Cellulari ed Ematologia - Divisione di Ematologia, Roma
  - Azienda Ospedaliera Universitaria Policlinico Tor Vergata, Rome

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: GIMEMA Foundation Website — http://www.gimema.it